CLINICAL TRIAL: NCT06599333
Title: Effectiveness of Digital Marketing Strategies to Improve Adherence to Chronic Medications: The e-MedAL Study
Brief Title: Effectiveness of Digital Marketing Strategies to Improve Adherence to Chronic Medications
Acronym: e-MedAL
Status: Completed | Type: Observational
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Georges Hatem, Associate Clinical and Epidemiological Professor, Lebanese University
Other Study IDs: 18/24/D
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Adherence to Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients coming to community pharmacies and taking at least the same medication for 6 months
  Interventions: Behavioral: Adherence to Care

INTERVENTIONS:
Behavioral: Adherence to Care — Questionnaire to assess the perception and readiness of patients in Lebanon towards the effectiveness of digital marketing strategies to improve their adherence to medications they take chronically
  The following sections will be considered:
  * General Characteristics of the Participants
  * Medical and medication history
  * Assessment of adherence to chronic medications (Likert scale)
  * Digital Marketing Strategies to improve adherence to chronic medications (Likert scale)
  * Perceived barriers to adopting digital marketing strategies in Lebanon (Likert scale)

SUMMARY:
In the Middle East, particularly Lebanon, the adoption of digital health interventions has been growing. Mobile health (mHealth) platforms, social media campaigns, and telemedicine services are being integrated into healthcare systems. However, while digital marketing for health promotion is gaining traction globally, few studies have specifically examined its impact on medication adherence in Lebanon. The e-MedAL Study aims to fill this gap by evaluating whether tailored digital marketing strategies can foster better adherence among patients with chronic diseases, taking into account the local healthcare infrastructure and cultural context. Lebanon faces unique challenges in managing chronic diseases due to its healthcare system, which is fragmented and highly privatized. The ongoing economic crisis, coupled with the COVID-19 pandemic, has placed additional stress on healthcare delivery, making it difficult for patients to maintain consistent access to medications. Moreover, the high cost of chronic medications, coupled with the population's general reliance on out-of-pocket expenditures, contributes to non-adherence.

Exploring cost-effective and scalable interventions like digital marketing becomes vital in this context. Lebanon has a high internet and mobile phone penetration rate, which presents an opportunity for leveraging digital tools to promote health. By utilizing culturally tailored messaging and communication strategies, the e-MedAL Study has the potential to improve medication adherence rates significantly. This, in turn, would alleviate the burden on healthcare resources, enhance patient outcomes, and reduce the economic impact of poorly managed chronic diseases in the country. Furthermore, the success of this initiative could serve as a model for other countries in the region facing similar healthcare challenges. Lebanon's diverse and tech-savvy population makes it an ideal test case for assessing the role of digital marketing in healthcare, particularly in resource-constrained settings.

DETAILED DESCRIPTION:
The study focuses on the role of digital marketing in improving medication adherence for chronic diseases in Lebanon. Here's a detailed breakdown of the study:

1. Study Overview and Purpose Chronic diseases like diabetes, hypertension, and cardiovascular disorders are growing global health concerns. One of the biggest challenges is ensuring long-term adherence to prescribed treatments, which, if not followed, leads to poor health outcomes and higher healthcare costs .

   The e-MedAL study investigates how digital marketing strategies-such as mobile applications, social media campaigns, and online education-can improve medication adherence among patients in Lebanon . It evaluates the local healthcare infrastructure and cultural factors affecting adherence.
2. State of Digital Marketing in Healthcare Digital marketing has revolutionized how healthcare providers engage with patients. By offering more personalized and interactive communication channels, it provides opportunities to boost medication adherence. Digital tools like reminders, educational campaigns, and behavioral nudges have been shown to improve adherence by as much as 17% across various chronic diseases .

   Lebanon's high internet penetration presents an opportunity to implement these strategies. However, the country also faces unique challenges, such as a fragmented healthcare system, economic difficulties, and a reliance on out-of-pocket payments, making adherence a significant issue .
3. Research Format and Methodology (PECO) Population: Patients residing in Lebanon who have been taking chronic medications for at least six months.

   Exposure: The use of digital marketing strategies to improve medication adherence.

   Comparison: A questionnaire-based assessment to evaluate patients' perceptions and readiness to adopt digital marketing strategies.

   Outcomes: Correlation between the effectiveness of digital strategies and patient adherence, along with demographic characteristics.
4. Questionnaire Sections General Characteristics: Participants provide demographic information such as age, education, smoking habits, and economic status .

   Medical and Medication History: Participants detail their chronic conditions, medication routines, and healthcare provider preferences .

   Adherence Assessment: Using a Likert scale, participants assess how closely they follow their prescribed medication regimen .

   Effectiveness of Digital Marketing: This section assesses how digital reminders, educational content, social media, and telemedicine services influence medication adherence .

   Perceived Barriers: Participants indicate potential challenges in using digital health tools, such as internet access, privacy concerns, and trust in digital channels .
5. Study Timeline and Outcome The study began on July 15th, 2024, and is ongoing (IRB Faculty of Pharmacy, Lebanese University).

The expected outcomes include a thesis, a scientific publication, and possibly a presentation at an international conference .

The study aims to provide insights that could serve as a model for other countries facing similar healthcare challenges, particularly in resource-constrained settings like Lebanon.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking the same medication for at least six months
* Lebanese patients
* Those who agree to participate in the study

Exclusion Criteria:

* Those with electronic illiteracy
* Those who are not themselves responsible for purchasing the medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the general population residing in Lebanon and taking the same medication for at least six consecutive months
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of digital marketing strategies | through study completion, an average of 3 months
  Correlation between the score of the schemes, in addition to some inter-item correlation assessment, as mentioned earlier, and the participants general characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Hatem, Principal Investigator — Lebanese University
Locations (1):
- Lebanese University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided